CLINICAL TRIAL: NCT07311525
Title: Efficacy of Ultrasound-guided Retro Superior Costotransverse Ligament Space Block Versus External Oblique Intercostal Plane Block for Postoperative Analgesia in Laparoscopic Sleeve Gastrectomy: A Prospective Randomized Study
Brief Title: Ultrasound-Guided RSCTL vs EOIP Block for Analgesia in Sleeve Gastrectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Dina Mahmoud Fakhry, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Management, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FMBSUREC/05102025/Fakhry
Record Dates: First submitted 2025-12-10; First posted 2025-12-31 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Patient Satisfaction
Keywords: Sleeve Gastrectomy; Postoperative Analgesia; External Oblique Intercostal Plane Block; Retro superior costotransverse ligament space block
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- retro-SCTL block (Active Comparator): Participants in the (group retro-SCTL) will receive ultrasound-guided retro-SCTL space block after intubation. Following hydrodissection with 2 ml of 0.9% saline to confirm the correct needle tip position, 20 ml 0.25% bupivacaine was injected. The same procedure was then repeated with 20 ml 0.25% bupivacaine on the contralateral side.
  Interventions: Procedure: ultrasound-guided Retro superior costotransverse ligament space block
- EOI block (Active Comparator): Participants in the (group EOI) will receive ultrasound-guided EOI block after intubation. Following hydrodissection with 2 ml of 0.9% saline to confirm the correct needle tip position, 20 ml 0.25% bupivacaine was injected. The same procedure was then repeated with 20 ml 0.25% bupivacaine on the contralateral side.
  Interventions: Procedure: ultrasound-guided External Oblique Intercostal Plane Block

INTERVENTIONS:
Procedure: ultrasound-guided Retro superior costotransverse ligament space block — Participants will receive ultrasound-guided Retro superior costotransverse ligament space block after intubation. Following hydrodissection with 2 ml of 0.9% saline to confirm the correct needle tip position, 20 ml 0.25% bupivacaine was injected. The same procedure was then repeated with 20 ml 0.25% bupivacaine on the contralateral side.
  Arms: retro-SCTL block
Procedure: ultrasound-guided External Oblique Intercostal Plane Block — Participants will receive ultrasound-guided External Oblique Intercostal Plane Block after intubation.Following hydrodissection with 2 ml of 0.9% saline to confirm the correct needle tip position, 20 ml 0.25% bupivacaine was injected. The same procedure was then repeated with 20 ml 0.25% bupivacaine on the contralateral side.
  Arms: EOI block

SUMMARY:
The aim of this study is to compare the effect of ultrasound-guided retro-SCTL space block and EOI block on opioid consumption within 24 hours after LSG.

DETAILED DESCRIPTION:
Obesity is ranked as the 5th cause of preventable death and is associated with certain diseases, e.g., type 2 diabetes mellitus, hypertension, ischemic heart disease, hyperlipidemia, and sleep apnea. Egypt has the world's 18th highest obesity prevalence, according to the World Health Organization (WHO). Bariatric surgery is the most effective treatment for weight loss, reducing obesity-related comorbidities and mortality. This surgery has been shown to improve quality of life. Bariatric surgery is now universally performed laparoscopically and is the most performed elective surgery in patients with morbid obesity. Laparoscopic sleeve gastrectomy (LSG) has been shown to be related to lower complication rates, shorter hospital stays, and earlier re-engagement in normal activities than open procedures. However, postoperative pain is common. Pain often originates from port sites in the abdominal wall. As LSG requires removal of the relatively large resected gastric segment, this often requires enlargement of the trocar site and the fascial incision, which adds to the pain. Postoperative pain may be significant and has a negative impact on recovery, respiration, hemodynamics, mentation, ambulation, bowel function, and length of hospital stay. Also, opioid analgesia in obese patients is associated with serious adverse effects such as hypopnoea, hypoxaemia, drowsiness, ileus, vomiting, delayed ambulation, and mortality. These complications are compounded by pre-existing obstructive sleep apnea (OSA), cardiorespiratory insufficiency, psychiatric disorders, and chronic opioid use, which may be present in obese patients. Although epidural anesthesia is effective in pain control, positioning is extremely difficult in obese patients. Some regional anesthesia techniques such as transverse abdominis plane (TAP) block, quadratus lumborum (QL) block, and erector spinae plane (ESP) block may be used as a part of a multimodal analgesic regimen to reduce opioid consumption

. However, technical challenges such as difficulty in identifying the structures and limitations in needle movement may be experienced due to the deep anatomical location of structures when performing these blocks in patients with obesity.

Intertransverse process block (ITPB) is a paraspinal thoracic nerve block technique where the local anesthetic (LA) is injected into the thoracic "intertransverse tissue complex", behind the superior costotransverse ligament (SCTL). The retro superior costotransverse ligament space (retro-SCTL space) block is a novel ITPB, targeting the fat-filled space in the retro-SCTL space. ITPB may be technically simpler and safer to avoid pleural puncture than a thoracic paravertebral block (TPVB) since it does not require direct needle access to the thoracic paravertebral space.

External oblique intercostal plane (EOI) block, a nerve block , has an efficacy range of T6-10. EOI block is one of the novel interfascial plane blocks. EOI block can be performed as part of multimodal analgesia for upper abdominal surgeries. In addition, easy visualization of the application area with ultrasound guidance is an advantage for obese patients. While both retro-SCTL and EOI blocks are emerging techniques, a direct comparison of their analgesic efficacy and opioid-sparing effects in the context of LSG has not yet been performed. This study aims to directly address this gap.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 to 65 years
* Both genders
* American Society of Anesthesiologists (ASA) physical status I-II
* Body mass index (BMI) > 40 kg m-2,

Exclusion Criteria:

* Obesity secondary to an endocrine disorder
* known allergic diathesis to any drugs used in the study
* Presence of serious systemic illness (e.g., severe cardiac, pulmonary, renal, or hepatic dysfunction),
* Coagulation dysfunction
* Pre-existing psychological disorders
* Current use of analgesic or psychotropic medications
* Infection at a potential injection site
* Ahistory of chronic pain
* Conversion to laparotomy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
cumulative morphine consumption within the first 24 hours. | 24 hours post operative
  cumulative morphine consumption within the first 24 hours.

SECONDARY OUTCOMES:
Visual analogue scale (VAS) score for pain | 30 minutes, 1, 3, 6, 12, 24 hours postoperatively
  The VAS is a pain rating scale. Scores are based onself-reported measures of symptoms that are recorded witha single handwritten mark placed at one point along thelength of a 10-cm line that represents a continuum betweenthe two ends of the scale-"no pain" on the left end (0 cm) ofthe scale and the "worst pain" on the right end of the scale(10 cm).Visual analogue scale (VAS) score: will be assessed at rest and during movement at 30 min, 1, 3, 6, 12, 24 h postoperatively. A score ≤ 3 will be considered acceptable for pain relief. Supplementary rescue analgesia will be administered in the form of morphine IV 2 mg (at VAS ≥ 4), which may be repeated after 20 minutes.
A Sedation scale | Initial 24 hours postoperatively
  A Sedation scale will be applied to determine the sedation scores (0 = awake, 1 = drowsy, 2 = asleep but arousable, and 3 = deeply asleep). A sedation score of > 0 indicates being sedated at any time throughout the initial postoperative 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Dina M Fakhry, MD, Principal Investigator — Beni-Suef University
Locations (1):
- Beni-Suef University hospital, Banī Suwayf, Beni Suweif Governorate, Egypt